CLINICAL TRIAL: NCT02000141
Title: The Australian Colonic Advanced Mucosal Neoplasia and Endoscopic Resection Study - a Prospective Observational Cohort Study
Brief Title: The Australian Colonic Advanced Mucosal Neoplasia and Endoscopic Resection Study
Acronym: ACER/AMN
Status: Active, not recruiting | Type: Observational
Sponsor: Professor Michael Bourke (Other)
Responsible Party: Sponsor-Investigator, Professor Michael Bourke, Director of Gastrointestinal Endoscopy, Western Sydney Local Health District
Organization: Western Sydney Local Health District (Other)
Other Study IDs: HREC2013/8/4.5(3778); AU RED HREC/13/WMEAD/233 (Other: WSLHD HREC Ethics Committee)
Record Dates: First submitted 2013-11-26; First posted 2013-12-03 (Estimated); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Colonic Polyps
MeSH Terms: conditions — Colonic Polyps | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Endoscopic Mucosal Resection: Endoscopic Mucosal Resection of Colonic Advanced Mucosal Lesions
  Interventions: Procedure: Endoscopic Mucosal Resection

INTERVENTIONS:
Procedure: Endoscopic Mucosal Resection

SUMMARY:
To enhance understanding of the risk factors for AMN, improve lesion assessment and prediction of submucosal invasive cancer, improve endoscopic resection efficacy, reduce complications of WF-EMR and improve the understanding of the progression of large lesions to cancer

DETAILED DESCRIPTION:
The Australian Colonic Endoscopic Mucosal Resection study (ACE), is a multicentre prospective observational study which examined WF-EMR of colonic AMN (Ethics approval No. HREC JH/TG 2008/9/6.1(2858)). This project now has an extensive dataset from 8 leading colonic endoscopic resection centres in Australia on more than 1500 lesions resected over 4 years since June 2008.

The ACE study has been successful in addressing several aspects of the resection of AMN, resulting in several high profile papers in internationally recognised journals. The collection of this data has produced robust information on the efficacy of the procedure4, recurrence rates7, bleeding complications8 and mortality when compared to surgery5. Single centre analysis of the ACE dataset at Westmead has also allowed insights into how to refine the procedure to improve outcomes. The target sign is now a recognised indication for the placement of clips to prevent perforation9, CO2 insufflation for WF-EMR has been shown to be superior to air insufflation10 and succinylated gelatin (Gelofusine®) has been shown to be superior to normal saline as a submucosal lifting agent11.

There remain a number of unanswered questions regarding the endoscopic resection of large sessile lesions and expanding the ACE dataset in a new cohort of patients will allow these to be addressed. Enhancing the prediction of submucosal invasive cancer, advanced lesion classification, refinement of the assessment of deep injury, submucosal injectate constituents, the optimum electrosurgical resection methods, prevention and prophylaxis of bleeding, and subtype analyses of the different histological groups comprising AMN will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for endoscopic resection of a large sessile colonic polyp or laterally spreading tumour ≥20mm in size.
* Age > 18 years
* Able to give informed consent to involvement in the clinical study

Exclusion Criteria:

• Unable to provide informed consent for involvement

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to a study centre for colonic WF-EMR of a known sessile colonic polyp or laterally spreading tumour (LST) ≥20mm in size.
Sampling Method: Non-Probability Sample
Enrollment: 1281 (Actual)
Dates: Start 2014-01; Primary Completion 2017-01 (Actual); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence | 6-60 months
  Follow up colonoscopies as per standard of care for 6 - 60 months noting and treating any recurrence.

SECONDARY OUTCOMES:
Cancer prediction | Initial procedure
  By properly assessing the lesion it is hoped that we will be able to provide the greater Gastroenterology community with a tool which can be used to properly identify benign and cancerous lesions to decrease the number of benign lesions being referred to surgery.
Improved Endoscopic Resection | 0-60 months
  By assessing the lesion at resection and following up with standard of care colonoscopies it is anticipated that there will be an improved endoscopic resection efficacy therefore reducing the risk of recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bourke, MBBS, Principal Investigator — South West Sydney Area Health Service
Locations (1):
- Westmead Endoscopy Unit, Westmead, New South Wales, Australia

REFERENCES:
- [Derived] Gauci JL, Mandarino FV, Kerrison C, Whitfield AM, O'Sullivan T, Gupta S, Lam B, Perananthan V, Cronin O, Lee EY, Williams SJ, Burgess N, Bourke MJ. Margin thermal ablation eliminates size as a risk factor for recurrence after piecemeal endoscopic mucosal resection of large non-pedunculated colorectal polyps. Gut. 2025 Apr 7;74(5):752-760. doi: 10.1136/gutjnl-2024-333563. PMID 40044497
- [Derived] Gauci JL, Whitfield A, Medas R, Kerrison C, Mandarino FV, Gibson D, O'Sullivan T, Cronin O, Gupta S, Lam B, Perananthan V, Hourigan L, Zanati S, Singh R, Raftopoulos S, Moss A, Brown G, Klein A, Desomer L, Tate DJ, Williams SJ, Lee EY, Burgess N, Bourke MJ. Prevalence of Endoscopically Curable Low-Risk Cancer Among Large (>/=20 mm) Nonpedunculated Polyps in the Right Colon. Clin Gastroenterol Hepatol. 2025 Mar;23(4):555-563.e1. doi: 10.1016/j.cgh.2024.07.017. Epub 2024 Jul 31. PMID 39089517
- [Derived] Tate DJ, Vosko S, Bar-Yishay I, Desomer L, Shahidi N, Sidhu M, McLeod D, Bourke MJ. Incomplete mucosal layer excision during EMR: a potential source of recurrent adenoma (with video). Gastrointest Endosc. 2024 Sep;100(3):501-509. doi: 10.1016/j.gie.2024.01.030. Epub 2024 Jan 25. PMID 38280532
- [Derived] Tate DJ, Desomer L, Argenziano ME, Mahajan N, Sidhu M, Vosko S, Shahidi N, Lee E, Williams SJ, Burgess NG, Bourke MJ. Treatment of adenoma recurrence after endoscopic mucosal resection. Gut. 2023 Oct;72(10):1875-1886. doi: 10.1136/gutjnl-2023-330300. Epub 2023 Jul 6. PMID 37414440
- [Derived] O'Sullivan T, Tate D, Sidhu M, Gupta S, Elhindi J, Byth K, Cronin O, Whitfield A, Craciun A, Singh R, Brown G, Raftopoulos S, Hourigan L, Moss A, Klein A, Heitman S, Williams S, Lee E, Burgess NG, Bourke MJ. The Surface Morphology of Large Nonpedunculated Colonic Polyps Predicts Synchronous Large Lesions. Clin Gastroenterol Hepatol. 2023 Aug;21(9):2270-2277.e1. doi: 10.1016/j.cgh.2023.01.034. Epub 2023 Feb 12. PMID 36787836
- [Derived] Cronin O, Sidhu M, Shahidi N, Gupta S, O'Sullivan T, Whitfield A, Wang H, Kumar P, Hourigan LF, Byth K, Burgess NG, Bourke MJ. Comparison of the morphology and histopathology of large nonpedunculated colorectal polyps in the rectum and colon: implications for endoscopic treatment. Gastrointest Endosc. 2022 Jul;96(1):118-124. doi: 10.1016/j.gie.2022.02.022. Epub 2022 Feb 24. PMID 35219724
- [Derived] Shaleve Y, Sabo E, Bourke MJ, Klein A. Computerized image analysis of blood vessels within mucosal defects for the prediction of delayed bleeding following colonic endoscopic mucosal resection: a pilot study. Endoscopy. 2021 Aug;53(8):837-841. doi: 10.1055/a-1258-8992. Epub 2020 Nov 10. PMID 32898919
- [Derived] Bahin FF, Heitman SJ, Rasouli KN, Mahajan H, McLeod D, Lee EYT, Williams SJ, Bourke MJ. Wide-field endoscopic mucosal resection versus endoscopic submucosal dissection for laterally spreading colorectal lesions: a cost-effectiveness analysis. Gut. 2018 Nov;67(11):1965-1973. doi: 10.1136/gutjnl-2017-313823. Epub 2017 Oct 7. PMID 28988198
- [Derived] Burgess NG, Hourigan LF, Zanati SA, Brown GJ, Singh R, Williams SJ, Raftopoulos SC, Ormonde D, Moss A, Byth K, Mahajan H, McLeod D, Bourke MJ. Risk Stratification for Covert Invasive Cancer Among Patients Referred for Colonic Endoscopic Mucosal Resection: A Large Multicenter Cohort. Gastroenterology. 2017 Sep;153(3):732-742.e1. doi: 10.1053/j.gastro.2017.05.047. Epub 2017 Jun 2. PMID 28583826
- [Derived] Burgess NG, Bassan MS, McLeod D, Williams SJ, Byth K, Bourke MJ. Deep mural injury and perforation after colonic endoscopic mucosal resection: a new classification and analysis of risk factors. Gut. 2017 Oct;66(10):1779-1789. doi: 10.1136/gutjnl-2015-309848. Epub 2016 Jul 27. PMID 27464708